CLINICAL TRIAL: NCT05522764
Title: Predictors of Infective Endocarditis Among Patients Managed for Staphylococcus Aureus Bacteremia, Particularly Staphylococcus Aureus Bacteriuria, and Time to Blood Culture Positivity
Acronym: BACT_URIE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: BACT_URIE
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Bacteremia; Endocarditis, Bacterial
MeSH Terms: conditions — Bacteremia; Endocarditis, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Staphylococcus aureus is a frequent cause of primary or secondary bacteremia. It is also responsible for many cases of infective endocarditis, for which the therapeutic management is specific. The frequency of infective endocarditis among Staphylococcus aureus bacteremias varies between 2.7% and 23.4%. Many factors associated with the risk of developing endocarditis in patients with S. aureus bacteremia have been described. Two parameters of potential interest remain excluded from this work: blood culture growth time, a marker of bacterial inoculum, and the presence of bacteriuria, which is common during bacteremia. The objective of this study is to evaluate the interest of these two parameters in the prediction of the presence of endocarditis during S. aureus bacteremia. Investigators will conduct a retrospective study including all patients managed for Staphylococcus aureus bacteremia and in whom a urine culture was performed.

The primary objective is to describe the factors associated with the occurrence of endocarditis in patients managed for S. aureus bacteremia and who received a urine cytobacteriological examination (UCE).

The secondary objectives are: to evaluate the factors associated with the occurrence of S. aureus bacteriuria in patients with S. aureus bacteremia and to evaluate the risk factors for mortality in patients managed for S. aureus bacteremia.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age for whom:

  * Blood cultures returned positive for S. aureus
  * A cytobacteriological examination of the urine was performed concomitantly with the positive blood culture for S. aureus
  * Has been tested for infective endocarditis by echocardiography.
* French-speaking patient

Exclusion Criteria:

* Patient with S. aureus bacteremia who has not had an ECBU or echocardiography performed
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his or her data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age for whom blood cultures returned positive for S. aureus and a cytobacteriological examination of the urine was performed concomitantly with the positive blood culture for S. aureus, have been tested for infective endocarditis by echocardiography.
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Factors associated with the occurrence of endocarditis | Month 1
  This outcome corresponds to the description of predictive factors for infective endocarditis in patients with S. aureus bacteremia.

SECONDARY OUTCOMES:
Factors associated with the occurrence of S. aureus bacteriuria | Month 1
  This outcome corresponds to the comparison of patients with S. aureus bacteremia and same-germ bacteriuria to those without same-germ bacteriuria.
Risk factors for mortality | Month 1
  This outcome corresponds to the comparison of patients who died in the setting of their S. aureus bacteremia to surviving patients.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit PILMIS, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Al Mohajer M, Darouiche RO. Staphylococcus aureus Bacteriuria: Source, Clinical Relevance, and Management. Curr Infect Dis Rep. 2012 Dec;14(6):601-6. doi: 10.1007/s11908-012-0290-4. PMID 22945379
- [Background] Chang FY, Peacock JE Jr, Musher DM, Triplett P, MacDonald BB, Mylotte JM, O'Donnell A, Wagener MM, Yu VL. Staphylococcus aureus bacteremia: recurrence and the impact of antibiotic treatment in a prospective multicenter study. Medicine (Baltimore). 2003 Sep;82(5):333-9. doi: 10.1097/01.md.0000091184.93122.09. PMID 14530782
- [Background] Le Moing V, Alla F, Doco-Lecompte T, Delahaye F, Piroth L, Chirouze C, Tattevin P, Lavigne JP, Erpelding ML, Hoen B, Vandenesch F, Duval X; VIRSTA study group. Staphylococcus aureus Bloodstream Infection and Endocarditis--A Prospective Cohort Study. PLoS One. 2015 May 28;10(5):e0127385. doi: 10.1371/journal.pone.0127385. eCollection 2015. PMID 26020939
- [Background] Thwaites GE, Edgeworth JD, Gkrania-Klotsas E, Kirby A, Tilley R, Torok ME, Walker S, Wertheim HF, Wilson P, Llewelyn MJ; UK Clinical Infection Research Group. Clinical management of Staphylococcus aureus bacteraemia. Lancet Infect Dis. 2011 Mar;11(3):208-22. doi: 10.1016/S1473-3099(10)70285-1. PMID 21371655
- [Background] Tubiana S, Duval X, Alla F, Selton-Suty C, Tattevin P, Delahaye F, Piroth L, Chirouze C, Lavigne JP, Erpelding ML, Hoen B, Vandenesch F, Iung B, Le Moing V; VIRSTA/AEPEI Study Group. The VIRSTA score, a prediction score to estimate risk of infective endocarditis and determine priority for echocardiography in patients with Staphylococcus aureus bacteremia. J Infect. 2016 May;72(5):544-53. doi: 10.1016/j.jinf.2016.02.003. Epub 2016 Feb 22. PMID 26916042
- [Background] Abu Saleh O, Fida M, Asbury K, Narichania A, Sotello D, Bosch W, Vikram HR, Palraj R, Lahr B, Baddour LM, Sohail MR. Prospective Validation of PREDICT and Its Impact on the Transesophageal Echocardiography Use in Management of Staphylococcus aureus Bacteremia. Clin Infect Dis. 2021 Oct 5;73(7):e1745-e1753. doi: 10.1093/cid/ciaa844. PMID 32569366
- [Background] Horino T, Sato F, Hosaka Y, Hoshina T, Tamura K, Nakaharai K, Kato T, Nakazawa Y, Yoshida M, Hori S. Predictive factors for metastatic infection in patients with bacteremia caused by methicillin-sensitive Staphylococcus aureus. Am J Med Sci. 2015 Jan;349(1):24-8. doi: 10.1097/MAJ.0000000000000350. PMID 25250988
- [Background] Kaasch AJ, Fowler VG Jr, Rieg S, Peyerl-Hoffmann G, Birkholz H, Hellmich M, Kern WV, Seifert H. Use of a simple criteria set for guiding echocardiography in nosocomial Staphylococcus aureus bacteremia. Clin Infect Dis. 2011 Jul 1;53(1):1-9. doi: 10.1093/cid/cir320. PMID 21653295
- [Background] Huggan PJ, Murdoch DR, Gallagher K, Chambers ST. Concomitant Staphylococcus aureus bacteriuria is associated with poor clinical outcome in adults with S. aureus bacteraemia. J Hosp Infect. 2008 Aug;69(4):345-9. doi: 10.1016/j.jhin.2008.04.027. Epub 2008 Jul 3. PMID 18602184
- [Background] Kahn F, Resman F, Bergmark S, Filiptsev P, Nilson B, Gilje P, Rasmussen M. Time to blood culture positivity in Staphylococcus aureus bacteraemia to determine risk of infective endocarditis. Clin Microbiol Infect. 2021 Sep;27(9):1345.e7-1345.e12. doi: 10.1016/j.cmi.2020.11.007. Epub 2020 Nov 13. PMID 33197608